CLINICAL TRIAL: NCT06214312
Title: Pulmonary Ultrasound for the Assessment of Atelectasis in Anesthetized Children Using a Laryngeal Mask Airway: a Randomized Double-Blinded Controlled Trial That Compares Spontaneous and Pressure Support Ventilation
Brief Title: Pulmonary Ultrasound for the Assessment of Atelectasis in Anesthetized Children Using a Laryngeal Mask Airway.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: B0762023231006
Record Dates: First submitted 2023-12-04; First posted 2024-01-19 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-01

CONDITIONS: Atelectasis; Hypoxemia
Keywords: lung ultrasounds; laryngeal mask airway; anesthetized children; spontaneous ventilation; pressure support ventilation; positive end expiratory pressure
MeSH Terms: conditions — Pulmonary Atelectasis; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Spontaneous ventilation: Anesthetized Children ventilated with a laryngeal mask airway in spontaneous ventilation with a positive end expiratory pressure of 5cmH2O.
  Interventions: Diagnostic Test: Lung Ultrasounds
- Pressure support ventilation: Anesthetized Children ventilated with a laryngeal mask airway in pressure support ventilation with a positive end expiratory pressure of 5cmH2O, maximum pressure not exceeding 15cmH2O.
  Interventions: Diagnostic Test: Lung Ultrasounds

INTERVENTIONS:
Diagnostic Test: Lung Ultrasounds — An ultrasound exam of the lungs to identify possible areas of atelectasis.

SUMMARY:
This study will use lung ultrasounds (LUS) to evaluate the incidence and severity of intraoperative atelectasis in anesthetized children undergoing minor surgery using a laryngeal mask airway. The children will be randomly assigned to be left in spontaneous ventilation with a Positive End Expiratory Pressure (PEEP) of 5cmH2O or to be ventilated with a pressure support mode.

DETAILED DESCRIPTION:
It is well known and described the deleterious effect that general anesthesia (GA) has on functional residual capacity (FRC), especially in children. This population is at higher risk of decreasing FRC during GA because of their lower capacity for elastic retraction and lower relaxation volume comparing to adults, predisposing them to the development of atelectasis and airway closure. These factors will lead to intrapulmonary shunts, which may impair the gas exchange and consequently oxygenation. By reducing the intrapulmonary shunt, Positive End Expiratory Pressure (PEEP) during controlled mechanical ventilation in patients with healthy lungs optimizes the FRC. However, the available data for an optimal ventilation strategy, including optimal PEEP, using a laryngeal mask airway (LMA) in the pediatric population are scarce, even though this device is frequently used in all age groups for brief general anesthesia.

Diagnosing anesthesia-induced atelectasis in the perioperative period can be possible by using lung ultrasounds (LUS), a simple, easily accessible, non-invasive and radiation free technique, which might help determine the impact in pulmonary aeration between different ventilation strategies. In our study, we will focus on comparing spontaneous ventilation (VS) with a PEEP of 5 cmH2O and pressure-support ventilation using a LMA in anesthetized children undergoing minor and elective outpatient surgery.

ELIGIBILITY:
Inclusion Criteria:

* fasted children between 12 months and 8 years of age; American Society of Anesthesiology (ASA) score I or II without lung disease; baseline pulse oximetry in room air >96%; scheduled for minor urological surgery (circumcision) under general anesthesia; written parent's agreement.

Exclusion Criteria:

* ASA score > II, chronic lung disease, airway infection in the last 15 days, impossibility of insertion of LMA.

Ages: 1 Year to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 12 months and 8 years scheduled for minor urologic surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
Pulmonary aeration | during surgery and in the immediate postoperative period
  Compare the Lung Aeration Score in the two groups

SECONDARY OUTCOMES:
Plethysmography | during surgery and in the immediate postoperative period.
  Correlation between Lung Aeration Score and Plethysmography
Ventilatory parameters | during surgery
  Correlation between Lung Aeration Score and Ventilatory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Carini, MD, Principal Investigator — Resident in Anesthesiology
Locations (1):
- Chu St. Pierre, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376
- [Background] Acosta CM, Lopez Vargas MP, Oropel F, Valente L, Ricci L, Natal M, Suarez Sipmann F, Tusman G. Prevention of atelectasis by continuous positive airway pressure in anaesthetised children: A randomised controlled study. Eur J Anaesthesiol. 2021 Jan;38(1):41-48. doi: 10.1097/EJA.0000000000001351. PMID 33009190
- [Background] Fiedler MO, Schatzle E, Contzen M, Gernoth C, Weiss C, Walter T, Viergutz T, Kalenka A. Evaluation of Different Positive End-Expiratory Pressures Using Supreme Airway Laryngeal Mask during Minor Surgical Procedures in Children. Medicina (Kaunas). 2020 Oct 21;56(10):551. doi: 10.3390/medicina56100551. PMID 33096743
- [Background] Joshi P, Vasishta A, Gupta M. Ultrasound of the pediatric chest. Br J Radiol. 2019 Aug;92(1100):20190058. doi: 10.1259/bjr.20190058. Epub 2019 May 16. PMID 31095416
- [Background] Templeton TW, Hoke LK, Yaung J, Aschenbrenner CA, Rose DM, Templeton LB, Bryan YF. Comparing 3 ventilation modalities by measuring several respiratory parameters using the ProSeal laryngeal mask airway in children. J Clin Anesth. 2016 Nov;34:272-8. doi: 10.1016/j.jclinane.2016.04.031. Epub 2016 May 15. PMID 27687391
- [Background] Lim B, Pawar D, Ng O. Pressure support ventilation vs spontaneous ventilation via ProSeal laryngeal mask airway in pediatric patients undergoing ambulatory surgery: a randomized controlled trial. Paediatr Anaesth. 2012 Apr;22(4):360-4. doi: 10.1111/j.1460-9592.2012.03819.x. PMID 22380745
- [Background] von Goedecke A, Brimacombe J, Keller C, Hoermann C, Loeckinger A, Rieder J, Kleinsasser A. Positive pressure versus pressure support ventilation at different levels of PEEP using the ProSeal laryngeal mask airway. Anaesth Intensive Care. 2004 Dec;32(6):804-8. doi: 10.1177/0310057X0403200612. PMID 15648991